CLINICAL TRIAL: NCT04012203
Title: Temporal Relationship in Recovery of Sensory, Motor and Tissue Variables in an Experimental Exercise-induced Muscle Pain Model of the Wrist Extensor Muscles
Brief Title: Multivariable Recovery After Exercise-induced Muscle Pain in the Forearm Muscles
Status: Completed | Type: Observational
Sponsor: Universidad San Jorge (Other)
Responsible Party: Sponsor
Other Study IDs: PI18/385
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Musculoskeletal Pain; Healthy; Delayed Onset Muscle Soreness
Keywords: Musculoskeletal pain; Delayed Onset Muscle Soreness; Pain mechanisms; Pressure Pain Threshold; Myotonometer; Maximal isometric strength; Manual dexterity
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy subjects: Participants free from any pain specific to the upper limb during the past 3 months, chronic pain or other disease.

SUMMARY:
This study investigates the evolution of sensory, motor and tissue variables following exercise-induced pain in wrist extensor muscles in healthy subjects.

DETAILED DESCRIPTION:
The aim of this study is to determine how is the normalization process of sensory (pressure pain thresholds, subjective pain sensation, self-recovery perception), motor (maximal isometric strength, active range of motion, manual dexterity) and tissue (myotonometer) variables after an experimental pain model in the extensor forearms muscles, by delayed onset muscle soreness after an eccentric exercise in healthy subjects. This way will be possible to establish 1) if there are differences in the time of normalization for each variable; 2) if there is a correlation between each variable and self-recovery perception.

Seven assessment sessions are performed in a 14-days period. Day 0 (baseline assessment 1), Day 7 (baseline assessment 2, pre exercise), Day 7 (post exercise), Day 8 (24-hours post exercise), Day 9 (48-hours post exercise), Day 10 (72-hours post exercise), Day 14 (1-week post exercise).

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy subjects of both sexes.
* Age: 18-50.
* Being free from any pain specific to the upper limb and/or in general.

Exclusion Criteria:

* History of acute or chronic painful condition in the previous 3 months.
* Regular medication intake for any reason.
* History of severe injury in the upper extremity (e.i. fracture).
* Prior surgery in the upper limb.
* Diagnosed of any chronic pain syndrome (fibromyalgia, migraine, etc.) or severe disease.

Withdrawal Criteria:

* Being involved in new physical stimulus, which volunteer is not used to.
* Micronutrient supplementation intake.
* NSAIDs or other medication intake.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young-adults free of pain or disease and without history of severe injury.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Changes in Pressure Pain Thresholds: pressure algometry | Day-1 (baseline assessment 1), Day-7 (baseline assessment 2, pre exercise), Day-7 (post-exercise), Day-8 (24 hours post-exercise), Day-9 (48 hours post-exercise), Day-10 (72 hours post-exercise), Day-14 (1-week post-exercise).
  Changes in pressure pain thresholds will be determined with pressure algometry bilaterally over the forearm, leg and shoulder. Pressure Pain Threshold is defined as the exact time point where the pressure is first being perceived at painful.
Changes in subjective perception of pain and recovery: Likert Scale | Day-1 (baseline assessment 1), Day-7 (baseline assessment 2, pre exercise), Day-7 (post-exercise), Day-8 (24 hours post-exercise), Day-9 (48 hours post-exercise), Day-10 (72 hours post-exercise), Day-14 (1-week post-exercise).
  A modified 7-item Likert Scale for pain ("0" No pain - "6" Severely disabling pain) and a visual analogue scale (0-10 cm) for self-recovery perception will be filled up to show subjective perception along the follow-up period.

SECONDARY OUTCOMES:
Changes in mechanical properties of the muscle | Day-1 (baseline assessment 1), Day-7 (baseline assessment 2, pre exercise), Day-7 (post-exercise), Day-8 (24 hours post-exercise), Day-9 (48 hours post-exercise), Day-10 (72 hours post-exercise), Day-14 (1-week post-exercise).
  Changes in mechanical properties of the muscle will be determined with myotonometer bilaterally over the forearm.
Changes in manual dexterity | Day-1 (baseline assessment 1), Day-7 (baseline assessment 2, pre exercise), Day-7 (post-exercise), Day-8 (24 hours post-exercise), Day-9 (48 hours post-exercise), Day-10 (72 hours post-exercise), Day-14 (1-week post-exercise).
  Changes in manual dexterity of both upper limbs will be assessed by the Nine Hole Peg Test. Participants will had to place 9 pegs in a specifically designed board as fast as possible.
Changes in maximal isometric force | Day-1 (baseline assessment 1), Day-7 (baseline assessment 2, pre exercise), Day-7 (post-exercise), Day-8 (24 hours post-exercise), Day-9 (48 hours post-exercise), Day-10 (72 hours post-exercise), Day-14 (1-week post-exercise).
  Changes in wrist extensors maximal isometric strength will be assessed with hand-held dynamometry.
Changes in active range of motion | Day-1 (baseline assessment 1), Day-7 (baseline assessment 2, pre exercise), Day-7 (post-exercise), Day-8 (24 hours post-exercise), Day-9 (48 hours post-exercise), Day-10 (72 hours post-exercise), Day-14 (1-week post-exercise).
  Changes in active range of motion of the wrist will be assessed in both sides using a digital inclinometer.
Level of catastrophizing | Day-1 (baseline), Day-14 (1-week post-exercise).
  Punctuation obtained in Pain Catastrophizing Scale (PCS). It comprises 13 items which focus on thoughts and feelings encountered while experiencing pain. Each item is scored from 0 (not at all) to 4 (all the time) with a total PCS score range from 0-52 points, where higher scores indicating higher levels of pain catastrophizing.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad San Jorge, Villanueva de Gállego, Zaragoza, Spain